CLINICAL TRIAL: NCT04090463
Title: A Phase II Study of Primary Chemotherapy, Stereotactic Body Radiation Therapy, and Intraoperative Radiation Therapy in Borderline Resectable Pancreatic Adenocarcinoma
Brief Title: IORT on Borderline Resectable Pancreatic Cancer
Acronym: PancFORT
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Logistic and financial reasons
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Salvatore Paiella, MD, Principal Investigator, Universita di Verona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PancFORT
Record Dates: First submitted 2019-09-10; First posted 2019-09-16 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Borderline Resectable Pancreatic Cancer
Keywords: Pancreatic cancer; Borderline resectable pancreatic cancer; Intraoperative radiotherapy (IORT); Total neoadjuvant therapy
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IORT group (Experimental): Intraoperative administration of 10 to 20 Gy after surgery or as an "in situ" treatment in case resection will not be performed
  Interventions: Radiation: Intraoperative radiotherapy

INTERVENTIONS:
Radiation: Intraoperative radiotherapy — IORT will be delivered as follows:
  1. Radical resection --> delivery of 10-15 Gy to the tumor bed
  2. Non radical resection --> delivery of 15-20 Gy to the tumor "in situ"

SUMMARY:
This phase II study investigates the efficacy of IORT for patients with borderline resectable pancreatic cancer. The purpose of the study is to investigate whether the addition of IORT, after FOLOFIRINOX-base chemotherapy, and SBRT, increases the 3-year survival rate. A total of 101 patients will be enrolled, and these patients will receive IORT of 10 to 20 Gy, according to the resection status (to the tumor bed after resection, or to the tumor in situ in case of non-resection).

DETAILED DESCRIPTION:
Treatment outcomes of borderline resectable pancreatic cancer are still poor even after completion of FOLFIRINOX-based chemotherapy and radical resection. A growing body of literature is demonstrating that Stereotactic body radiation therapy (SBRT) and Intraoperative radiotherapy (IORT), within a multimodal approach, allow to obtain better oncological outcome, at the price of low to negligible rates of morbidity and mortality. The investigators hypothesize that a "total neoadjuvant" scenario, with the best current therapy, based on up to 6 months of FOLFIRINOX (minimum 4), SBRT and IORT (in situ or after surgery) would increase the disease-specific survival of borderline resectable pancreatic cancer patients. An historical cohort will be used as a comparison group.

Considering the intention-to-treat design and the institutional rates of chemotherapy completion and exploration/resection of borderline resection pancreatic cancer patients, a total of 100 patients will be enrolled in this phase II trial. Patients submitted to IORT, will receive IORT of 10 to 20 Gy according to the resection status (to the tumor bed after resection, or to the tumor in situ in case of non-resection).

ELIGIBILITY:
Inclusion Criteria:

* • Biopsy-proven, previously untreated borderline resectable PC, defined according to the NCCN guidelines v1.2019;

  * Age 18-80 years;
  * Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1;
  * Adequate bone marrow function (absolute neutrophil count ≥1500 per cubic millimeter; platelet count ≥100.000 per cubic millimeter; hemoglobin level ≥10 g per deciliter), liver function (serum total bilirubin level ≤1.5 times the upper limit of the normal range), and renal function (creatinine clearance ≥50 ml per minute);
  * Ability to understand the characteristics of the clinical trial;
  * Written informed consent.

Exclusion Criteria:

* • Ampullary, biliary, or duodenal adenocarcinoma; pancreatic adenocarcinoma in the background of an intraductal papillary mucinous neoplasia (IPMN), other uncommon pancreatic adenocarcinomas (acinar-cell, squamous, giant-cell osteoclastic-like);

  * Invasive cancer in the last 5 years requiring radiation therapy to the upper abdomen or chemotherapy;
  * Symptomatic heart failure or coronary artery disease;
  * Pregnant or lactating women;
  * Impaired mental state or language problems.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Disease-specific survival | 36 months

SECONDARY OUTCOMES:
Progression-free survival | 36 months
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 36 months
Rate of margin-free surgery | 30 days
Rate of surgical complications | Up to 90 days after surgery
Resection rate | Intraoperative

CONTACTS AND LOCATIONS:
Locations (1):
- General and Pancreatic Surgery Unit, Pancreas Institute, University of Verona Hospital, Verona, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Palta M, Willett C, Czito B. The role of intraoperative radiation therapy in patients with pancreatic cancer. Semin Radiat Oncol. 2014 Apr;24(2):126-31. doi: 10.1016/j.semradonc.2013.11.004. PMID 24635869
- [Result] Krempien R, Roeder F. Intraoperative radiation therapy (IORT) in pancreatic cancer. Radiat Oncol. 2017 Jan 10;12(1):8. doi: 10.1186/s13014-016-0753-0. PMID 28069018
- [Result] Cai S, Hong TS, Goldberg SI, Fernandez-del Castillo C, Thayer SP, Ferrone CR, Ryan DP, Blaszkowsky LS, Kwak EL, Willett CG, Lillemoe KD, Warshaw AL, Wo JY. Updated long-term outcomes and prognostic factors for patients with unresectable locally advanced pancreatic cancer treated with intraoperative radiotherapy at the Massachusetts General Hospital, 1978 to 2010. Cancer. 2013 Dec 1;119(23):4196-204. doi: 10.1002/cncr.28329. Epub 2013 Sep 4. PMID 24006012
- [Result] Murphy JE, Wo JY, Ryan DP, Jiang W, Yeap BY, Drapek LC, Blaszkowsky LS, Kwak EL, Allen JN, Clark JW, Faris JE, Zhu AX, Goyal L, Lillemoe KD, DeLaney TF, Fernandez-Del Castillo C, Ferrone CR, Hong TS. Total Neoadjuvant Therapy With FOLFIRINOX Followed by Individualized Chemoradiotherapy for Borderline Resectable Pancreatic Adenocarcinoma: A Phase 2 Clinical Trial. JAMA Oncol. 2018 Jul 1;4(7):963-969. doi: 10.1001/jamaoncol.2018.0329. PMID 29800971
- [Derived] Paiella S, Malleo G, Simoni N, Micera R, Guariglia S, Cavedon C, Marchegiani G, Esposito A, Landoni L, Casetti L, Tuveri M, Milella M, Secchettin E, Manzini G, Bovo C, De Pastena M, Fontana M, Salvia R, Mazzarotto R, Bassi C. A phase II trial proposal of total neoadjuvant treatment with primary chemotherapy, stereotactic body radiation therapy, and intraoperative radiation therapy in borderline resectable pancreatic adenocarcinoma. BMC Cancer. 2021 Feb 16;21(1):165. doi: 10.1186/s12885-021-07877-7. PMID 33593311